CLINICAL TRIAL: NCT00639977
Title: Effect of Acupuncture on Intraocular Pressure
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Daniel Meira Freitas, Universidade Federal de São Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CEP 1196/07
Record Dates: First submitted 2008-03-14; First posted 2008-03-20 (Estimated); Last update posted 2008-03-20 (Estimated); Status verified 2008-03

CONDITIONS: Healthy
Keywords: Intraocular Pressure; Acupuncture; Healthy Volunteers
MeSH Terms: interventions — Acupuncture Therapy; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 2 (Sham Comparator): 20- minute session of acupuncture with needles inserted in false points allocated 1 cm from the true points in areas without acupuncture's meridians
  Interventions: Other: Sham
- 1 (Active Comparator): 20-minute session of acupuncture with needles inserted in specific points (Tong Zi Liao, Yang Bai and Jing Ming)
  Interventions: Other: Acupuncture
- 3 (No Intervention)

INTERVENTIONS:
Other: Acupuncture — 20-minute session of acupuncture with needles inserted in specific points: Tong Zi Liao, Yang Bai and Jing Ming
  Arms: 1
Other: Sham — 20- minute session of acupuncture with needles inserted in false points allocated 1 cm from the true points in areas without acupuncture's meridians
  Arms: 2

SUMMARY:
To evaluate the short-term effect of acupuncture on the intraocular pressure (IOP).

Methods: A randomized controlled trial. Healthy volunteers will be randomly allocated to three groups: Acupuncture group - will be submitted to a 20-minute session of acupuncture with needles inserted in specific points (Tong Zi Liao, Yang Bai and Jing Ming); Sham group - will be submitted to a 20- minute session of acupuncture with needles inserted in false points located 1 cm from true points in areas without acupuncture's meridians; and Control group - no intervention. IOP measurement by a masked investigator using Goldmann applanation tonometry immediately before the intervention, as well as 30 minutes and 24 hours after the acupuncture.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers

Exclusion Criteria:

* glaucoma
* past intraocular surgery
* corneal alterations
* medications that interferes with the intraocular pressure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-09; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
variation of the intraocular pressure | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Meira-Freitas, MD, Principal Investigator — Universidade Federal de São Paulo; Angelino J Cariello, MD, Study Chair — Universidade Federal de São Paulo; Luiz Alberto S Melo Jr., MD, Study Director — Universidade Federal de São Paulo
Locations (1):
- Departamento de Oftalmologia - UNIFESP, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Meira-Freitas D, Cariello AJ, Vita RC, Tabosa A, Melo LA Jr. Short-term effect of acupuncture on intraocular pressure in healthy subjects. Acupunct Med. 2010 Mar;28(1):25-7. doi: 10.1136/aim.2009.001081. PMID 20351373